CLINICAL TRIAL: NCT01389739
Title: Evaluation of a Multi-faceted Intervention to Improve Continuity of Care for Patients With Lung Cancer
Brief Title: Intervention to Improve Continuity of Care in Lung Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Michèle Aubin, Professeur, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 020097
Record Dates: First submitted 2011-02-14; First posted 2011-07-08 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2013-05

CONDITIONS: Lung Cancer
Keywords: continuity of care; interprofessional collaboration
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exposed to the intervention (Experimental): Patients in the intervention arm will be exposed to a multi-faceted intervention to improve continuity of care; the intervention includes 4 components: 1) systematic appointments with FP at 3-month interval during the study period; 2) transmission to FP of a standardized comprehensive summary before each appointment; 3)systematic transmission to the oncology team of patients' information resulting from FP visits; 4) development of a priority access to FP for cancer patients
  Interventions: Other: Multi-faceted intervention to improve continuity of care
- Usual care (No Intervention)

INTERVENTIONS:
Other: Multi-faceted intervention to improve continuity of care — Periodic exchange of information between FP and oncology team and systematic appointments with FP at 3-month interval
  Other Names: Change in practice organization
  Arms: Exposed to the intervention

SUMMARY:
Many authors have recognized the need to overcome the different barriers to continuity of cancer care, such as inadequate communication between specialists and family physicians (FP), insufficient information provided for the long-term follow-up care and difficulties to transfer back to FP the responsibility for cancer care at the end of treatments. This study aims to assess the effectiveness of a multi-faceted intervention to improve continuity of care for patients with lung cancer. Newly diagnosed lung cancer patients who have a FP will be randomly assigned to either the intervention group or to usual care and they will be followed at baseline, 3, 6, 9, 12, 15 and 18 months ( or until death for those with a survival of less than 18 months). The intervention comprises 4 components: 1) systematic appointments with FP at 3-month interval ; 2) transmission to FP of a standardized comprehensive summary before each appointment; 3) systematic transmission to the oncology team of patients' information resulting from FP visits; 4) development of a priority access to FP for cancer patients. In both groups, outcomes related to patients and to care processes will be measured at baseline and then after 3, 6, 9, 12, 15 and 18 months (or until death for those with a survival of less than 18months). Patients' principal family caregiver will be invited to participate to the study and they will complete questionnaires at baseline, at 6 months and at the end of the study. In addition, patients' FP will also be invited to complete a questionnaire at baseline and at the end of the study.

DETAILED DESCRIPTION:
Lung cancer patients from both the intervention and the control group will complete validated questionnaires at baseline and then after 3, 6, 9, 12, 15 and 18 months (or until death for those with a survival of less than 18months) to assess their perceived collaboration between their FP and the oncology team (from an adaptation of Nielsen et al.'s validated questionnaire (2003)), their quality of life (from the EORTC-QLQ-C30), pain and other symptom relief (from the EORTC-QLQ-LC13), their level of distress, anxiety and depression (from the HADS), their self-efficacy (from an adaptation of Lorig et al.'s validated questionnaire (1996)). Several processes of care will also be measured at the same intervals: number of exchanges of information, number of visits to FP, number of answered/unanswered calls from FP, delay to return patients' calls, responsibility for care by FP at the terminal phase of cancer, service utilization (ER visits, hospitalization, community health services). The investigators will also measure in patients' principal family caregivers, their perceived collaboration between FP and the oncology team (same questionnaire than the one used for patients but adapted to family caregivers), their distress (from the IDPESQ), psychological burden (from the CBS-EOLC) and self-efficacy (same questionnaire than the one used for patients but adapted to family caregivers . Finally, measures related to FP will include their perceived collaboration with the oncology team (same questionnaire than the one used for patients and family caregivers but adapted to FPs).

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed adult patients with lung cancer, with a prognosis of at least 3 months

Exclusion Criteria:

* cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2009-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Mean score of perceived collaboration between FP and the oncology team (from 0 to 100) | 18 months
  Adaptation of Nielsen et al.'s questionnaire used to measure collaboration between health professionals (2003)

SECONDARY OUTCOMES:
Mean score of Global Quality of life | 18 months
  EORTC-QLC-C30 and EORTC-QLQ-LC13 questionnaires
Mean score of Distress, Anxiety and Depression | 18 months
  HADS and IDPESQ questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Michele Aubin, MD, PhD, Principal Investigator — Laval University
Locations (1):
- Institut universitaire de cardiologie et pneumologie de Québec (IUCPQ), Québec, Quebec, Canada